CLINICAL TRIAL: NCT05995236
Title: Prostate-Specific Membrane Antigen (PSMA) Radionuclide Therapy for the Treatment of Metastatic Castration-Resistant Prostate Cancer
Brief Title: Prostate-Specific Membrane Antigen (PSMA) Radionuclide Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 019.NMD.2022.D
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: PSMA radionuclide therapy — Collect clinical data related to treatment of PSMA-positive metastatic castration-resistant prostate cancer treated with PSMA radionuclide therapy

SUMMARY:
This study is a single-center registry study collecting clinical data regarding the treatment of PSMA-positive metastatic castration-resistant prostate cancer treated with PSMA radionuclide therapy per the treating physician's discretion. Clinical data from candidates for or who undergo the PSMA procedure at Methodist Dallas Medical Center from August 2022 to August 2027 will be collected after discharge and patients will undergo clinical follow-up per the treating physician's discretion.

DETAILED DESCRIPTION:
This study is a single-center registry study collecting clinical data regarding the treatment of PSMA-positive metastatic castration-resistant prostate cancer treated with PSMA radionuclide therapy per the treating physician's discretion. Clinical data from candidates for or who undergo the PSMA procedure at Methodist Dallas Medical Center from August 2022 to August 2027 will be collected after discharge and patients will undergo clinical follow-up per the treating physician's discretion.

Participants will be followed for two years following the first PSMA procedure. During these visits, participants will also be asked to report any change in their medications. Participants will not need to visit the study doctor more often than their usual treatment unless they have other medical needs. However, if participants experience any significant change in their medical condition they may be asked to have additional tests such as computed tomography (CT) scans, blood tests, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1. >18 years of age
* 2. Diagnosed with PSMA-positive metastatic castration-resistant prostate cancer and - has consented to undergo PSMA nuclear therapy per the treating physician. Specifically:

  * Metastatic or Locally Advanced AND Inoperable
  * Clear disease progression on PSMA-PET/CT
  * PSMA-PET/CT scan positive disease within 6 weeks
  * Labs:

    * Hemoglobin: >8 g/dL
    * White blood cell count: >2K cells/µL
    * Platelet (Thrombocyte) count: >75 x 109/L
  * No prior therapy with Radium-223 Dichloride

Exclusion Criteria:

* Patients who do not meet the Inclusion Criteria laid out in section 4.2 will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The plan for Methodist Dallas Medical Center will be to collect data from 10-20 patients with PSMA-positive metastatic castration-resistant prostate cancer per year for anticipated 50-100 total patients over the next five years. We estimated this number based on the number of patient with prostate cancer treated within Methodist Heath System.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-08-02 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
collect clinical data related to treatment of PSMA-positive metastatic castration-resistant prostate cancer | Clinical data from candidates for or who undergo the PSMA procedure at Methodist Dallas Medical Center from August 2022 to August 2027 will be collected after discharge and patients will undergo clinical follow-up per the treating physician's discretion
  To collect clinical data related to patient characteristics, treatment responses and survival outcomes related to the treatment of PSMA-positive metastatic castration-resistant prostate cancer treated with PSMA radionuclide therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Bageac, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided